CLINICAL TRIAL: NCT01262131
Title: A Randomized, Double-blind, Placebo-controlled Evaluation of the Application of Magnetic Fields Using the Resonator Device for the Treatment of Fibromyalgia: Pilot Study Protocol
Brief Title: Evaluation of Magnetic Fields to Treat Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: Allen S. Braswell CEO, pico-tesla Magnetic Therapies, LLC, Pico-Tesla Magnetic Therapies, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10242-01
Record Dates: First submitted 2010-12-14; First posted 2010-12-17 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain associated with Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resonator Protocol A (Active Comparator)
  Interventions: Device: magnetic therapy protocol A
- Resonator Protocol B (Active Comparator): Application of magnetic fields using the Resonator device Protocol B
  Interventions: Device: magnetic therapy Protocol B
- Inactive Resonator (Placebo Comparator)
  Interventions: Device: placebo therapy

INTERVENTIONS:
Device: magnetic therapy protocol A — Application of magnetic fields using the Resonator device Protocol A
  Arms: Resonator Protocol A
Device: magnetic therapy Protocol B — Application of magnetic fields using the Resonator device Protocol B
  Arms: Resonator Protocol B
Device: placebo therapy — Application of inactive magnetic fields using the Resonator device
  Arms: Inactive Resonator

SUMMARY:
The purpose of this study is to see if a device called the Resonator can help to reduce pain and improve aspects of health and quality of life for people with fibromyalgia.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the efficacy of the Resonator device as an adjunctive therapy to reducing pain and improving aspects of health and quality of life that are relevant to individuals with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of fibromyalgia made by the study Principal Investigator (PI) according to the American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia.
* Rating of current Degree of Pain on the 0-10 Numeric Pain Intensity Scale of 4 or greater.
* Subject's use of pain relief medication(s) has been stable over the past 30 days, and subject is willing and able to maintain pre-existing use of pain relief medication(s) as his or her sole pain relief medication use, as needed, throughout study participation.
* Subject's use of insomnia medication(s) has been stable over the past 30 days, and subject is willing and able to maintain this existing use of insomnia medication(s) as his or her sole insomnia relief medication(s), as needed, throughout study participation.
* Subject has been on current (or no) medication regimen, unchanged for at least 30 days prior to study enrollment, and is willing and able to maintain that regular medication regimen, unchanged, throughout study participation.
* Willing and able to refrain from use of tender point injections throughout study participation.
* Willing and able to abstain from partaking in other/new treatments to improve fibromyalgia symptoms during study participation.
* Adequate contraceptive measures for female subjects. > 18 years of age or older.
* Male or female.

Exclusion Criteria:

* Any factors that might prevent the subject from completing a full course of therapy with the Resonator™ device, or from attending any of the scheduled study visits, or from completing any of the study measures.
* Subject suffers from co-existent chronic pain condition(s) of non-fibromyalgia origin, such as osteoarthritis, low back pain, neck pain, painful diabetic neuropathy and postherpetic neuropathic pain, that cannot be distinguished in severity and/or in type/sensation of pain from the pain originating from the subject's condition of fibromyalgia.
* Any other significant comorbidities that might impact the ability to evaluate the subject's satisfaction of the ACR 1990 Criteria for the Classification of Fibromyalgia, or for the subject to complete any of the study assessment tools.
* Tender point injections received within the prior one month.
* Current or past history of major psychiatric disturbance (e.g., schizophrenia, bipolar disorder, substance abuse).
* Known inflammatory rheumatic disease.
* Epilepsy/history of seizures/taking medication for epilepsy.
* HIV and other autoimmune disorders.
* Active cancer or treatment for cancer within last 6 months.
* Active infection(s).
* History of ECT
* Uncontrolled Hypertension.
* Advanced Pulmonary Disease.
* Unstable cardiac disease.
* Prosthetics or implants comprised of ferrous metals.
* Pacemakers, vagus nerve stimulators, or other functional electrical stimulators such as those commonly used for pain.
* Consumption of more than 21 alcoholic drinks per week.
* Pregnant, breast feeding, or planning pregnancy prior to end of study participation.
* Developmental disability or other cognitive impairment that would in the judgment of the PI impair adequate comprehension of the informed consent form or complete any of the study-related activities.
* Worker's compensation, receipt of disability or present/past litigation for monetary compensation pertaining to subject's fibromyalgia condition.
* Participation in other research within 30 days of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry I Jacobson, Ph.D, D.M.D., Principal Investigator

RESULTS

PARTICIPANT FLOW:
Groups:
- Resonator Protocol A: Application of magnetic fields using the Resonator device protocol A
- Resonator Protocol B: Application of magnetic fields using the Resonator device treatment protocol B
- Inactive Resonator: Application of inactive magnetic fields using the Resonator device
Period: Overall Study
Arm/Group | Resonator Protocol A | Resonator Protocol B | Inactive Resonator
Started | 5 | 4 | 4
Completed | 5 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resonator Protocol A | Resonator Protocol B | Inactive Resonator | Total
Number analyzed (Participants) | 5 | 4 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 4 | 13
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 13
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in 3-recording Average of the Subjects Daily Pain Rating on the 0-10 Numeric Pain Intensity Scale.
Description: Minimum scale value is '0' which represents 'no pain at all' and is the best outcome.
  Maximum scale value is '10 which represents the 'worst pain imaginable' and is the worse outcome.
Time Frame: 2 weeks (baseline to end of treatment)
Population: Analysis was by intention to treat which included all enrolled subjects in this case to study completion.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Resonator Protocol A | Resonator Protocol B | Inactive Resonator
Number analyzed (Participants) | 5 | 4 | 4
Scores on a scale | -3.69 (1.2) | -3.08 (1.2) | -1.97 (1)

ADVERSE EVENTS:
Arm/Group | Resonator Protocol A | Resonator Protocol B | Inactive Resonator
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes